CLINICAL TRIAL: NCT01321112
Title: Search for Transcriptional Biomarkers in a Conversion Protocol From Calcineurin Inhibitors to Mycophenolate Mofetil Monotherapy
Brief Title: Search for Transcriptional Biomarkers in a Conversion Protocol From Calcineurin Inhibitors to Mycophenolate Mofetil
Acronym: TBCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-071
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Gene Expression; Immunosuppression Conversion; Liver Transplantation
Keywords: Conversion; Mycophenolate mofetil; Calcineurin inhibitors; Liver transplantation; Gene expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conversion arm (Experimental): After screening procedure mycophenolate mofetil will be started (week -4) at a dose of 500 mg twice a day for two weeks and then (week -2) increased to 1000 mg twice a day and CNI will be reduced at the 50% of the initial dose. After two weeks (week 0) CNI will be completely discontinued (complete IS conversion). The investigators will follow up patients every 4 weeks up to 48 weeks after the complete IS conversion.
  Interventions: Drug: conversion from CNI to MMF

INTERVENTIONS:
Drug: conversion from CNI to MMF — After screening procedure mycophenolate mofetil will be started (week -4) at a dose of 500 mg twice a day for two weeks and then (week -2) increased to 1000 mg twice a day and CNI will be reduced at the 50% of the initial dose. After two weeks (week 0) CNI will be completely discontinued (complete IS conversion). The investigators will follow up patients every 4 weeks up to 48 weeks after the complete IS conversion.
  Other Names: Conversion

SUMMARY:
As is well known, immunosuppressive treatment (IS) after liver transplantation has several and frequents adverse effects that limit the survival of the graft and recipients. Because of that, it is desirable that these recipients were able to receive a mild IS regime with a better safety profile. An attempt to get that aim has been evaluated in several trials in the past, and consist in to change the IS regime from an calcineurin inhibitors (CNI) based to another less intense and with less adverse effects based on mycophenolate mofetil (MMF), which is known to have a better safety profile. The success rate of this strategy(i.e. complete conversion in absence of rejection) has a wide range from 100% to 50% approximately. However it is accepted that this strategy is associated with the improvement of several adverse effects of CNIs such as renal failure and dyslipemia. This study's aim is to perform IS conversion from CNI to MMF monotherapy and look for transcriptional biomarkers employing a whole genome expression study performed with microarrays at baseline on liver tissue and/or PBMCs to try to find a differential gene expression able to correlate with a successful conversion and thus, to generate a set of transcriptional biomarkers potentially able to predict the result of the IS conversion on an independent cohort of liver recipients.

DETAILED DESCRIPTION:
Introduction: Immunosuppressive treatment (IS) has several and frequents adverse effects; among them are: severe infections, diabetes mellitus, arterial hypertension, osteoporosis, neurologic disorders, renal failure, dyslipemias, increased cardiovascular risk, cancer, etc. After 5 years, 18% of liver receptors develop renal failure, the risk of developing cancer is three times higher after LT and 30% of liver graft receptors previously infected by hepatitis C virus (HCV) have cirrhosis 5 years after LT, probably because of the effect of IS on viral kinetics. An ideal situation would be that liver transplant recipients receive enough IS to inhibit the immune response against the allograft, while avoiding an excessive effect over the capacity of the immune system to recognize pathogens, tumoral cells and minimizing the adverse effects or even more, the indefinite graft acceptance in the complete absence of IS, concept that in clinic in called operational tolerance (OT). OT occurs in around 20% of liver recipients. So although the potential benefit is important it affects just a small fraction of liver recipients. A different but related strategy has been evaluated in several trials in the past, and consist in to change from an IS based on calcineurin inhibitors (CNI) to another less intense based on mofetil mycophenolate (MMF), which is known to have less adverse effects, preserve renal function and do not affect the function and proliferation of T regulatory cells, which are involved in the development of OT. In a recent study (in press), the investigators performed an IS withdrawal to over a hundred liver recipients and the investigators found that those who were classified as operationally tolerant (40%) where those with a longer time elapsed since LT to IS withdrawal, those who received lower doses of CNI and those who received MMF monotherapy. The investigators were able also to discriminate between operationally tolerant liver recipients and those who developed a rejection based on its differential gene expression (evaluated by whole genome microarray) just before the ISwithdrawal.

Study's aim: to perform IS conversion from CNI to MMF monotherapy and look for transcriptional biomarkers employing whole a genome expression study performed with microarrays at baseline on liver tissue and PBMCs to try to find a set differentially expressed genes able to correlate with a successful conversion and thus, to generate a set of transcriptional biomarkers potentially able to predict the result of the IS conversion on an independent cohort of liver recipients.

Methods: Forty patients will be recruited among our cohort of liver transplant recipients. The study will last 48 weeks. Inclusion criteria will be a) liver transplantation more than 2 years ago, b) stable graft function, b) no history of autoimmune liver disease, c) absence of rejection in the last 12 months, d) Use of calcineurin inhibitors (CNI) as monotherapy, e)absence of rejection on baseline liver biopsy, d) tacrolimus trough levels > 3 ng/ml or cyclosporine C2 levels > 30 ng/ml, e) signature of the informed consent form. After screening procedure mycophenolate mofetil will be started (week -4) at a dose of 500 mg twice a day for two weeks and then (week -2) increased to 1000 mg twice a day and CNI will be reduced at the 50% of the initial dose. After two weeks (week 0) CNI will be completely discontinued(complete IS conversion). The investigators will follow up patients every 4 weeks up to 48 weeks after the complete IS conversion. The complete study period will last 52 weeks. At baseline mRNA fron liver samples and peripheral blood mononuclear cells will be isolated. This mRNA will be used to evaluate whole genome expression using Affimetrix microarrays. Besides, T regulatory cells frequency will be measured using peripheral blood cell immunophenotyping at baseline and at the end of the follow up. Clinical variables will be evaluated to determined the evolution of renal function and other cardiovascular risk factors.

Expected results: The investigators expect that at the end of the study most of the recipients will have been able to have a successful rejection and a minor group (around 30%) will not be able to do it because of rejection. Then baseline mRNA samples will be used to perform whole genome microarrays. Using bioinformatics procedures the investigators will make an attempt to establish a differential gene expression among those with a successful conversion and those that develop rejection. This will allow the investigators to determine the smallest set of genes able to discriminate between those patients. Gene expression will be also correlated with peripheral blood cell immunophenotyping and clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation more than 2 years ago
* Stable graft function
* No history of autoimmune liver disease
* Absence of rejection in the last 12 months
* IS regime: calcineurin inhibitors (CNI) as monotherapy
* Absence of rejection in the baseline liver biopsy
* Signature of the informed consent form

Exclusion Criteria:

* total white cell count ≤ 2 x 109/L
* hemoglobin < 7.0 g/L
* platelet count ≤ 50x x 109/L
* systemic infection requiring therapy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of transcriptional biomarkers | 48 weeks
  Whole genome expresion study by microarrays will be use to determine the correlation between succesful conversion (yes/no) and the expression level of the most informative genes.

SECONDARY OUTCOMES:
Renal function improvement | 48 weeks
  20% of improvement on baseline serum creatinine compared to the serum creatinine at the end of the study.
Frequency of regulatory cells | 48 weeks
  The frequency of regulatory cells (CD4+FoxP3+ T cells) will be measured at baseline and at the end of the study.
Blood pressure | 48 weeks
  Reduction of baseline blood presure at the end of the study (48 weeks)
Total cholesterol reduction | 48 weeks
  Reduction of baseline serum cholesterol at the end of the study.
Uric acid reduction | 48 weeks
  Reduction of baseline uric acid serum level at the end of the study.
Reduction of glycosylated haemoglobin | 48 weeks
  Reduction of baseline glycosylated haemoglobin at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Benitez, MD, Principal Investigator — Gastroenterology Department. Pontificia Universidad Católica de Chile
Locations (1):
- Gastroenterology Department, Pontificia Universidad Catolica de Chile, Santiago, Santiago, RM, Chile

REFERENCES:
- [Background] Mells G, Neuberger J. Long-term care of the liver allograft recipient. Semin Liver Dis. 2009 Feb;29(1):102-20. doi: 10.1055/s-0029-1192059. Epub 2009 Feb 23. PMID 19235663
- [Background] Fishman JA. Infection in solid-organ transplant recipients. N Engl J Med. 2007 Dec 20;357(25):2601-14. doi: 10.1056/NEJMra064928. No abstract available. PMID 18094380
- [Background] Martinez-Llordella M, Lozano JJ, Puig-Pey I, Orlando G, Tisone G, Lerut J, Benitez C, Pons JA, Parrilla P, Ramirez P, Bruguera M, Rimola A, Sanchez-Fueyo A. Using transcriptional profiling to develop a diagnostic test of operational tolerance in liver transplant recipients. J Clin Invest. 2008 Aug;118(8):2845-57. doi: 10.1172/JCI35342. PMID 18654667
- [Background] Demirkiran A, Sewgobind VD, van der Weijde J, Kok A, Baan CC, Kwekkeboom J, Tilanus HW, Metselaar HJ, van der Laan LJ. Conversion from calcineurin inhibitor to mycophenolate mofetil-based immunosuppression changes the frequency and phenotype of CD4+FOXP3+ regulatory T cells. Transplantation. 2009 Apr 15;87(7):1062-8. doi: 10.1097/TP.0b013e31819d2032. PMID 19352129
- [Background] Farkas SA, Schnitzbauer AA, Kirchner G, Obed A, Banas B, Schlitt HJ. Calcineurin inhibitor minimization protocols in liver transplantation. Transpl Int. 2009 Jan;22(1):49-60. doi: 10.1111/j.1432-2277.2008.00796.x. PMID 19121146
- [Derived] Norero B, Serrano CA, Sanchez-Fueyo A, Duarte I, Torres J, Ocquetau M, Barrera F, Arrese M, Soza A, Benitez C. Conversion to mycophenolate mofetil monotherapy in liver recipients: Calcineurin inhibitor levels are key. Ann Hepatol. 2017 Jan-Feb 2017;16(1):94-106. doi: 10.5604/16652681.1226820. PMID 28051798